CLINICAL TRIAL: NCT01235208
Title: The Effect of a Low Carbohydrate Low Energy Ketogenic Diet Followed by Progressively Increased Intake of Low Glycemic Foods Over 7 Months on Weight and Body Composition and Hormonal Profile
Brief Title: The Effect of the Treatment Program "Dr. Fedon Lindbergs Vektcoach" on Body Weight and Composition and Hormonal Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eurodiet Scandinavia AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EDstudy
Record Dates: First submitted 2010-11-04; First posted 2010-11-05 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Overweight; Obesity; Metabolic Syndrome
Keywords: Overweight; Obesity; Metabolic syndrome; Diet; Carbohydrate; Low glycemic index; Eurodiet
MeSH Terms: conditions — Overweight; Obesity; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eurodiet treatment (Experimental)
  Interventions: Other: The "Dr. Fedon Lindbergs Vektcoach" Treatment

INTERVENTIONS:
Other: The "Dr. Fedon Lindbergs Vektcoach" Treatment — Diet and lifestyle treatment

SUMMARY:
The background for the trial is a number of previous studies indicating that it is especially important to restrict the intake of carbohydrates when treating overweight and metabolic diseases in general.

The purpose of the study is to obtain research data on the effects of an established treatment of overweight/obesity and its related metabolic disorders. The treatment, "Dr. Fedon Lindbergs Vektcoach", is a combination treatment where patients use low carbohydrate and low energy "Eurodiet" products in the initial phases. After the initial phases are completed, low glycemic normal foods are added to the diet until a sustainable and healthy diet is achieved. The treatment is of 7 month duration.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI)>35
* BMI>27 + one risk factor for cardiovascular disease or metabolic syndrome
* >18 years

Exclusion Criteria:

* Medicinal treatment of thyroid disease
* Pregnancy or planned pregnancy
* Taking of diet pills like Xenical or Sibutramine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Body weight/composition | 7 months

SECONDARY OUTCOMES:
Hormonal profile | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Pål T Jåbekk, M.Sc, Principal Investigator; Arne T Høstmark, Ph.D/Dr.Med, Study Director — Unaffiliated/ Study supervisor
Locations (1):
- Dr. Fedon Lindbergs Klinikk, Oslo, Norway